CLINICAL TRIAL: NCT03607682
Title: A Multi-Institutional Pilot Study of Prophylactic Cranial Tumor-Treating Fields for Patients With Extensive-stage Small Cell Lung Cancer
Brief Title: Tumor-Treating Fields Therapy in Preventing Brain Tumors in Participants With Extensive-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution and loss of funding
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Principal Investigator, Wade Iams, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 1747; NCI-2018-01428 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2018-07-11; First posted 2018-07-31 (Actual); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prevention (TTF therapy, NovoTTF-200A device) (Experimental)
  Interventions: Procedure: Tumor Treating Fields (TTF) Therapy; Device: NovoTTF-200A Device; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Tumor Treating Fields (TTF) Therapy — Undergo TTF therapy
Device: NovoTTF-200A Device — Undergo TTF therapy
Other: Quality-of-Life Assessment — Ancillary studies

SUMMARY:
This trial studies how well tumor-treating fields therapy works in preventing brain tumors in participants with small cell lung cancer that has spread to other places in the body. Tumor-treating fields therapy involves the use of the NovoTTF-200A which delivers alternating electrical fields, or tumor treating fields, through ceramic discs placed on the head. This electric force may slow and/or reverse tumor growth by disrupting the way cancer cells grow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the feasibility and compliance of NovoTTF-200A as prophylactic cranial tumor treatment fields (TTF) therapy, determined by percent (%) of patients continuing TTF therapy until intracranial tumor progression, discontinuation due to dose limiting toxicity (DLT), or 6 months.

SECONDARY OBJECTIVES:

I. To evaluate time to intracranial failure after NovoTTF-200A. II. To evaluate overall survival after NovoTTF-200A. III. To evaluate the rates of intracranial failure at 2, 4, 6, 8, 10, 12 months after NovoTTF-200A.

IV. To evaluate intracranial failure free survival after NovoTTF-200A. V. To evaluate the rate of decline in Hopkins Verbal Language Test-Revised (HVLT-R) free recall, delayed recall and delayed recognition, Controlled Oral Word Association Test (COWAT) and Trail Making Test (TMT) Parts A and B at 2, 4, 6, 8, 10, 12 months after NovoTTF-200A.

VI. To evaluate time to neurocognitive failure after NovoTTF-200A. VII. To evaluate neurocognitive failure-free survival after NovoTTF-200A. VIII. To evaluate quality of life using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC Quality of life Questionnaire C30) with BN20 addendum after NovoTTF-200A.

IX. To assess adverse events, severity, and frequency associated with NovoTTF-200A using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

OUTLINE:

Participants undergo tumor-treating fields therapy using the NovoTTF-200A device over 18 hours per day for a minimum of 4 weeks and up to 1 year in the absence of disease progression, unacceptable toxicity, or intracranial failure.

After completion of study treatment, participants are followed up at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of > 3 months
* Histologically proven extensive stage small cell lung carcinoma (ES-SCLC) (any T any N and any M stage) within 6 months prior to start of study treatment with the NovoTTF-200A, with a partial or complete response to at least four cycles of first-line chemotherapy
* Karnofsky performance status (KPS) > 70
* Neutrophil count > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L
* Bilirubin < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) < 2.5 x ULN or < 5 x ULN if patient has documented liver metastases
* Serum creatinine < 1.5 x ULN

Exclusion Criteria:

* Evidence of brain metastases on magnetic resonance imaging (MRI) of brain with and without contrast
* History of other prior malignancy within the past 5 years except for superficial skin cancers
* No severe comorbidities:

  * History of significant cardiovascular disease unless the disease is well controlled. Significant cardiac disease includes second/third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary activity results in fatigue, palpitation or dyspnea)
  * History of arrhythmia that is symptomatic or requires treatment. Patients with atrial fibrillation or flutter controlled by medication are not excluded from participation in the trial
  * History of cerebrovascular accident (CVA) within 6 months prior to start of study treatment
  * Active infection or serious underlying medical condition that would impair the ability of the patient to receive protocol therapy
  * History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent
* Active implantable electronic medical devices in the brain; a skull defect, a shunt, or bullet fragments
* Known allergies to medical adhesives or hydrogel
* Unable to operate the NovoTTF-200A device independently or with the help of a caregiver
* If a female, currently pregnant, breastfeeding, or unwilling to avoid pregnancy while on study treatment
* Concurrent brain directed therapy (beyond NovoTTF-200A as per protocol)
* Prior clinical trial participation with brain directed therapy
* Concurrent treatment clinical trials

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Attia, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was open to accrual from September 2018 to June 2020 at Vanderbilt Medical Center in Nashville, TN. Two participants were enrolled. The study stopped early due to loss of funding.
Pre-assignment Details: 2 participants were enrolled; 1 participant had disease progression and was not on the study long enough to be evaluable.
Period: Overall Study
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  Race: <=18 years | 0
  Race: Between 18 and 65 years | 1
  Race: >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Continuing Therapy Until Intracranial Tumor
Description: Count of patients developed intracranial tumor divided by total number of patients.
Time Frame: Up to 6 months
Population: patients on the therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Time to Intracranial Failure
Description: Time to intracranial failure with death as a competing risk will be estimated using cumulative incidence function (CIF) and reported with a one-sided 95% confidence interval.
Time Frame: Up to 3 years
Population: Data was not collected do to loss of funding.
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Population: Data was not collected do to loss of funding.
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Intracranial Failure
Description: Estimated using the cumulative incidence function
Time Frame: Up to 12 months
Population: Data was not collected do to loss of funding.
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 0

5. Secondary Outcome: Rate of Decline in Cognitive Function
Description: Measured by Hopkins Verbal Language Test
Time Frame: Up to 12 months
Population: Data was not collected do to loss of funding.
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Neurocognitive Failure
Description: Measured by Hopkins Verbal Language Test
Time Frame: Up to 3 years
Population: Data was not collected do to loss of funding.
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 0

7. Secondary Outcome: Neurocognitive Failure-free Survival
Description: Measured by Hopkins Verbal Language Test
Time Frame: Up to 3 years
Population: Data was not collected do to loss of funding.
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 0

8. Secondary Outcome: Evaluate Quality of Life Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30
Description: Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (scale 1-4)
Time Frame: Up to 3 years
Population: Data was not collected do to loss of funding.
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 0

9. Secondary Outcome: Incidence of Adverse Events
Description: Graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 12 months
Population: Patients on the therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: The adverse event reporting period began immediately following registration to treatment (start of use of the NovoTTF-200A device). Adverse events were collected for 8 weeks following treatment termination.
Arm/Group | Prevention (TTF Therapy, NovoTTF-200A Device)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT03607682/Prot_SAP_000.pdf